CLINICAL TRIAL: NCT00353613
Title: Prevention of Surgical Site Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Lillian Kao, Associate Professor - Surgery, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-050570; RWJ ID#57405
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Surgical Wound Infection
Keywords: Antibiotic prophylaxis
MeSH Terms: conditions — Surgical Wound Infection

ARMS (2):
- 1 (Other): LBJ Hospital
  Interventions: Behavioral: Package of targeted interventions to reduce error
- 2 (Other): Ben Taub Hospital
  Interventions: Behavioral: Package of targeted interventions to reduce error

INTERVENTIONS:
Behavioral: Package of targeted interventions to reduce error — Interventions will include changes in administration of antibiotics and the improved monitoring of blood glucose and body temperature peri-operatively.

SUMMARY:
The primary research question is whether interventions to prevent caregiver and system errors will increase the proportion of laparotomy patients who receive recommended measures to prevent surgical site infections.

DETAILED DESCRIPTION:
Background: Surgical site infections (SSIs) cause significant and largely preventable morbidity, mortality, and resource use due to failure to comply with evidence-based guidelines. Quality improvement programs report increased compliance with these guidelines, but are subject to a variety of biases.

Hypothesis: The primary hypothesis is that a targeted intervention program will increase the proportion of patients in a county hospital who receive recommended interventions to prevent SSIs, when assessed in the most rigorous feasible clinical trial. The specific aims of the trial are to establish practical surveillance measures to determine the percentage of patients whose care complies with 5 major guidelines to prevent SSIs; to use chart review, direct observation, attitude surveys, and focus groups to identify, quantify, and address latent and active errors linked to non-compliance, and to develop, implement, and assess the effectiveness of an intervention program to increase guideline compliance.

Study Design: An innovative trial design will be performed with 3 staggered phases in the two major county hospitals in Houston, TX. This design allows for adjustment for temporal trends and hospital differences in assessing the intervention program in a large, high-risk, disadvantaged urban population. Based on a compliance goal of 95%, this design has adequate power to detect even a small absolute increase ( >= 5%) above baseline in the percentage of patients receiving all 5 recommended preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparotomy at either Ben Taub Hospital or Lyndon Baines Johnson Hospital in Houston, Texas

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2007-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Proportion of laparotomy patients receiving recommended measures to prevent surgical site infections | 1 year

SECONDARY OUTCOMES:
Surgical site infections | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lillian S Kao, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas